CLINICAL TRIAL: NCT03465215
Title: Evaluation of Stricturing Crohn's Disease Using Digital Holographic Microscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-732-f-S
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Quantitative Phase Imaging

STUDY DESIGN:
Intervention Model Description: The investigators will include 29 CD patients with a symptomatic intestinal stricture requiring surgery. From these patients, the investigators will collect fullthickness surgical specimen from the non-stenotic and stenotic intestinal wall and will perform analysis using digital holographic microscopy and in histopathological analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of inflammation grade (Experimental): Tissue obtained by CD patients will be analyzed using digital holographic microscopy and comparing histological analysis.
  Interventions: Device: Digital holographic microscopy

INTERVENTIONS:
Device: Digital holographic microscopy — Tissue obtained from CD patients will be analyzed using digital holographic microscopy. Results will be compared between non-stenotic and stenotic tissue of the intestinal wall of CD patients.

SUMMARY:
Crohn's Disease (CD) patients, belonging to Inflammatory Bowel Disease (IBD), frequently suffer from uncontrolled intestinal inflammation. This can lead to severe disease complications requiring hospitalization. Up to 50% of all CD patients develope intestinal strictures. Intestinal strictures can be subdivided into predominantly inflammatory and predominantly fibrotic types. This subclassification in different types of strictures is important for clinical decision making: patients with predominantly fibrotic strictures would undergo surgery or interventional endoscopic treatment and patients with predominantly inflammatory strictures would be treated anti-inflammatory. To determining the degree of fibrosis and inflammation in CD strictures remains difficult.

Digital holographic microscopy (DHM) is a new imaging approach belonging to the group of quantitative phase imaging. DHM enables stain-free quantitative phase contrast imaging and provides the determination of an refractive index which directly correlated to tissue density.

This study aims to evaluate DHM for assessing the degree of fibrosis and inflammation in surgical specimen from patients with stricturing CD. The investigators collect full thickness surgical resection specimen from 29 patients with symptomatic CD strictures. More detailed, the investigators collect full thickness surgical resection specimen out of stenotic and non-stenotic bowel segments from each patient. For primary purposes, the investigators analyze the obtained tissue using DHM and compare differences of the refractive index, determined by DHM, between stenotic and non-stenotic parts of the intestinal wall. For secondary purposes, the investigators will correlate the findings made by DHM with a detailed analysis by a histopathologist using a scoring system (Goldstandard) to determine the degree of fibrosis and inflammation in the samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic intestinal Crohn's Disease stricture requiring surgery

Exclusion Criteria:

* Patients < 18 years
* Pregnancy
* Inability for an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the refractive index for characterising CD strictures | Directly after surgical resection, the investigators obtain fullthickness surgical specimen. Tissue will directly be transported to the laboratory. After processing, the tissue is ready for analysis and will be assessed within a period up to 90 weeks.
  Obtained intestinal tissue (non-stenotic and stenotic) tissue will be analyzed using digital holographic microscopy (DHM). DHM provides a refractive index which will be compared between non-stenotic and stenotic tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Bettenworth, Professor, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Unversity Clinic Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided